CLINICAL TRIAL: NCT01542385
Title: Immediate vs. Delayed Stenting After Primary Percutaneous Reperfusion in ST Elevation Myocardial Infarction
Brief Title: Primary Reperfusion Secondary Stenting Trial
Acronym: PRIMACY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Marc Jolicoeur, E. Marc Jolicoeur, MD MSc MHS FRCP-C FACC, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMACY
Record Dates: First submitted 2012-02-16; First posted 2012-03-02 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Delayed stenting; Deferred stenting; Late stenting; postponed stenting; Thrombectomy; Percutaneous coronary intervention; PCI; Angioplasty; STEMI; acute myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate stenting (Active Comparator): the stent selection (bare metal vs drug eluting) and implantation will be performed as recommended by current practice guidelines.
  Interventions: Procedure: Stent
- Delayed stenting (Experimental): participants randomised to delayed stenting will be treated with GPIIb-IIIa inhibitors for 12-18 hours after reperfusion followed by anticoagulation for until the control angiogram, expected no sooner than 18-24 hours after the index reperfusion.
  Interventions: Procedure: Stent

INTERVENTIONS:
Procedure: Stent — Percutaneous coronary intervention: reperfusion with a thrombectomy catheter or a small balloon angioplasty catheter, followed by coronary stenting
  Other Names: Thrombectomy catheter; Balloon angioplasty catheter; Coronary stent

SUMMARY:
The purpose of this research project is to improve how we treat heart attacks. The study will assess whether it might not be better to wait a few hours before implanting the coronary stent into the coronary artery rather than implanting it immediately, in order to allow the drugs to completely dissolve the clot. This might help to reduce the risks of the clot migrating and damaging the heart. By delaying coronary stent implantation, we hope to be able to reduce the size of the infarction and reduce the risk of suffering from heart failure following a heart attack.

DETAILED DESCRIPTION:
The PRIMACY trial seeks to assess whether a strategy of delayed stent implantation combined with adjunctive anticoagulation is superior to immediate stent implantation at improving cardiovascular outcomes in patients with mechanically reperfused ST-elevation Myocardial Infarction (STEMI). The investigators hypothesize that delayed stent implantation combined with systemic anticoagulation and maximal antiplatelet therapy will reduce the combined occurrence of cardiac death, non-fatal myocardial infarction, congestive heart failure, or unplanned target vessel revascularization over a 9-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years;
2. STEMI, presenting within 12 hours of symptoms onset, and persisting for more than 20 minutes;
3. ECG that fulfills any of the following criteria: ≥ 2 mm ST elevation in two anterior or lateral leads; or ≥ 1 mm ST elevation in two inferior leads; or new left bundle branch block (LBBB) with at least 1 mm concordant ST elevation;
4. Infarct-related artery with TIMI flow 0 or 1 at baseline angiogram;
5. Successful reperfusion (TIMI 2-3 flow), either spontaneously or after wire passage, thrombectomy, small size (≤ 2.0mm) angioplasty catheter, and persisting for more than 10 minutes;
6. Infarct related artery with a diameter above 2.5 mm.

Exclusion Criteria:

1. Prior STEMI in the qualifying coronary artery;
2. Coronary dissection following reperfusion;
3. STEMI caused by acute stent thrombosis or a venous or arterial bypass graft occlusion;
4. Significant left main disease, as determined by angiography (≥ 50%) or other imaging technologies;
5. Cardiac condition requiring emergent or urgent surgical repair;
6. Failed thrombolysis and rescue PCI;
7. High risk of bleeding;
8. Contraindication to either ticagrelor or GpIIb/IIIa inhibitors;
9. STEMI with Killip III-IV or cardiogenic shock or presenting as sudden death, ventricular fibrillation, or sustained ventricular tachycardia;
10. Women who are pregnant or breastfeeding;
11. Creatinine clearance < 20 ml/min;
12. Other contraindication to PCI;
13. Participation with another investigational drug or investigational device study within 30 days prior to randomization (participation to registries is allowed);
14. Any condition that in the opinion of the investigator would preclude compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2014-04; Primary Completion 2018-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The combined occurence of cardiac death, non-fatal myocardial infarction, congestive heart failure, and urgent target vessel revascularization | 9 months
  As defined by standardized definitions

SECONDARY OUTCOMES:
Major bleeding | 9 months
  As defined by the Bleeding Academic Research Consortium (BARC).

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Jolicoeur, MD MSc MHS, Study Chair — Montreal Heart Institute, Université de Montréal; Nandini Dendukuri, PhD, Study Director — Centre for Outcomes Research, McGill University Health Centre - Research Institute; Loic Belle, MD, Study Director — Hospital of Annecy, Centre Hospitalier Annecy Genevois, Annecy, France
Locations (16):
- Canada (5):
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM-Hôtel-Dieu de Montréal, Montreal, Quebec
  - Hôpital du Sacré Cœur de Montréal, Montreal, Quebec
  - Centre Hospitalier Régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - CHR CSSS de Trois Rivières, Trois-Rivières, Quebec
- France (11):
  - CH de Bastia, Bastia
  - CH de Cannes, Cannes
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Louis-Pasteur, Le Coudray
  - HCL Hopital Croix Rousse, Lyon
  - CH Annecy Genevois, Metz-Tessy
  - Ch de Montpellier-Hôpital A. de Villneuve, Montpellier
  - CH de Nimes, Nîmes
  - CH de Pau, Pau
  - CHU de Toulouse-Hôpital Rangueil, Toulouse
  - CH de Vichy, Vichy